CLINICAL TRIAL: NCT01860222
Title: A Prospective Randomized Trial of Surgical Resection Versus Percutaneous Local Ablative Therapy for Hepatocellular Carcinoma Complicating Clinically Significant Portal Hypertension Within the Milan Criteria
Brief Title: Surgical Resection Versus Percutaneous Local Ablative Therapy for Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospital, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EHBHKY2012-002-12
Record Dates: First submitted 2013-05-15; First posted 2013-05-22 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma With CSPH
Keywords: Hepatocellular carcinoma; CSPH; Hepatectomy; percutaneous local ablative; therapy (PLAT); randomized controlled trials(RCTs)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SR (Active Comparator)
  Interventions: Procedure: SR
- PLAT (Experimental)
  Interventions: Procedure: PLAT

INTERVENTIONS:
Procedure: SR
  Arms: SR
Procedure: PLAT
  Arms: PLAT

SUMMARY:
The aim of this study is to compare the operative complication and short-/long-term therapeutic effects of percutaneous local ablative therapy (PLAT) versus surgical resection(SR) on small hepatocellular carcinoma(HCC) patients with clinically significant portal hypertension(CSPH) so as to lend clinical and theoretical basis of the therapeutic schemes for the disease.

DETAILED DESCRIPTION:
HCC is a major health problem worldwide, with an estimated incidence ranging between 500,000 and 1,000,000 new cases annually. It is the fifth most common cancer in the world and the third most common cause of cancer-related death,especially in East-Asia countries.SR remains the first therapeutic option for a cure but is suitable only for 9%-27% of patients.The presence of significant background cirrhosis often precludes liver resection for HCC.Even though these HCC patients undergo SR，the incidence of posthepatectomy liver failure(PHLF) and death would be high，especially to HCC patients complicating CSPH，whose corresponding risk of PHLF and persistent PHLF were 59.02%and 14.75%respectively in our past study. It is extremely urgent to search a safe and effective means in this subgroup of HCC patients.PLAT, a recently developed local ablative technique, has attracted the greatest interest and popularity because of its effectiveness and safety,with a 3-year survival rate of 62-77%,a low treatment complication rate of 8-9% and a low treatment mortality rate of 0-0.5%.However, there is still debate on whether PLAT or SR is the most suitable therapy for HCC.To our knowledge,there have been no study on the therapy of HCC complicating CSPH.

ELIGIBILITY:
Inclusion Criteria:

1. 18 Years < ge ≤ 70 Y,KPS ≥ 70
2. A solitary HCC ≤ 5cm in diameter,or multiple HCC(≤3) ,each ≤3cm in diameter without evidence of radiologically definable vascular invasion or extrahepatic metastasis. allowing to both SR and PLAT
3. Child-Pugh class A or B,without history of encephalopathy,ascites refractory to diuretics,or variceal bleeding
4. NO previous treatment of HCC
5. Platelet count>40,000/mm3；prothrombin time prolongation of no more than 3 seconds
6. Patients who can understand this trial and have signed information consent

Exclusion Criteria:

1. metastatic liver cancer
2. Patients with apparent cardiac,pulmonary,cerebral and renal dysfunction,which may affect the treatment of HCC

3) Patients with other diseases which may affect the treatment mentioned

4） Patients participating in other clinical trials

5） Patients with a medical history of other malignant tumors

6) Pregnant and breast-feeding women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3 years

SECONDARY OUTCOMES:
local tumor progression | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, China